CLINICAL TRIAL: NCT05336591
Title: COVID-19, Obesity and Lifestyle in Children - Role of Professionals
Acronym: COLC-Pro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-1634
Record Dates: First submitted 2022-04-19; First posted 2022-04-20 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: COVID-19; COVID-19 Pandemic; Childhood Obesity; Overweight, Childhood
MeSH Terms: conditions — COVID-19; Pediatric Obesity | interventions — Pandemic Preparedness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Medical doctor
  Interventions: Other: Covid-19 pandemic
- Nurses (Pediatric department and youth healthcare)
  Interventions: Other: Covid-19 pandemic
- Other professionals in treatment (e.g. dieticians, physiotherapists)
  Interventions: Other: Covid-19 pandemic
- Other (such as policy makers)
  Interventions: Other: Covid-19 pandemic

INTERVENTIONS:
Other: Covid-19 pandemic — All participants worked during the Covid-19 pandemic in the preventive or curative healthcare for children with overweight and obesity. We will ask all professionals about their experiences during and after the pandemic.

SUMMARY:
In this study it is researched how preventive and curative healthcare for children with overweight and obesity was conducted during the Covid-19 pandemic, which barriers were noticed by professionals, and how new methods (such as e-health and telemonitorning) for coaching, communication and healthcare were used and experienced.

ELIGIBILITY:
Inclusion Criteria:

* Worked during the Covid-19 pandemic
* Works with children with overweight and / or obesity
* Works in The Netherlands

Exclusion Criteria:

* No knowledge of the Dutch language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Professionals working with children with overweight and/or obesity.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
Views and experiences of health care professionals working with children with overweight and obesity during the COVID-19 pandemic | 2 years after the start of the Covid-19 pandemic
  Views and experiences of health care professionals working with children with overweight and obesity during the COVID-19 pandemic measured with a questionnaire using open-end and closed-end (likert-scale) questions.
User experience | 2 years after the start of the Covid-19 pandemic
  User experience of professionals using ehealth options in healthcare for children with overweight or obesity, measured with a questionnaire using closed end and open end questions.

SECONDARY OUTCOMES:
Experiences | 2 years after the start of the Covid-19 pandemic
  In case more in-depth data is needed after the inital questionnaire, semi-structured interviews will be conducted to experiences of health care professionals during the Covid-19 pandemic.

CONTACTS AND LOCATIONS:
Overall Officials: Anita CE Vreugdenhil, Prof, Principal Investigator — MUMC+, Maastricht University
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided